CLINICAL TRIAL: NCT05564403
Title: FOLFOX in Combination With Binimetinib as 2nd Line Therapy for Patients With Advanced Biliary Tract Cancers With MAPK Pathway Alterations: A ComboMATCH Treatment Trial
Brief Title: Study of Chemotherapy, With or Without Binimetinib in Advanced Biliary Tract Cancers in 2nd Line Setting (A ComboMATCH Treatment Trial)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2022-07833; NCI-2022-07833 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY191-A6 (Other: Alliance for Clinical Trials in Oncology); EAY191-A6 (Other: CTEP); U10CA180821 (NIH)
Record Dates: First submitted 2022-09-27; First posted 2022-10-03 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Advanced Biliary Tract Carcinoma; Advanced Gallbladder Carcinoma; Advanced Intrahepatic Cholangiocarcinoma; Recurrent Biliary Tract Carcinoma; Recurrent Gallbladder Carcinoma; Recurrent Intrahepatic Cholangiocarcinoma; Stage III Distal Bile Duct Cancer AJCC v8; Stage III Gallbladder Cancer AJCC v8; Stage III Hilar Cholangiocarcinoma AJCC v8; Stage III Intrahepatic Cholangiocarcinoma AJCC v8; Stage IV Distal Bile Duct Cancer AJCC v8; Stage IV Gallbladder Cancer AJCC v8; Stage IV Hilar Cholangiocarcinoma AJCC v8; Stage IV Intrahepatic Cholangiocarcinoma AJCC v8; Unresectable Biliary Tract Carcinoma; Unresectable Gallbladder Carcinoma; Unresectable Intrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Gallbladder Neoplasms; Cholangiocarcinoma; Klatskin Tumor | interventions — binimetinib; Biopsy; Specimen Handling; Fluorouracil; dehydroftorafur; Leucovorin; Magnetic Resonance Spectroscopy; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (mFOLFOX6) (Active Comparator): Patients receive leucovorin IV over 2 hours and oxaliplatin IV over 2 hours on day 1, and fluorouracil IV over 46-48 hours on days 1-2. Cycles repeat every 14 days in the absence of disease progression or unacceptable toxicity. Patients undergo collection of blood during screening and on study, and undergo CT with contrast, MRI, or FDG-PET throughout the trial as clinically indicated. Patients may also undergo bone scans on study and may undergo biopsies throughout the study as clinically indicated.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Fluorouracil; Drug: Leucovorin Calcium; Procedure: Magnetic Resonance Imaging; Drug: Oxaliplatin
- Arm 2 (binimetinib, mFOLFOX6) (Experimental): Patients receive binimetinib PO on days 1-14, and leucovorin IV, oxaliplatin IV, and fluorouracil IV as in Arm 1. Cycles repeat every 14 days in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO or MUGA and collection of blood during screening and on study, and undergo CT with contrast, MRI, or FDG-PET throughout the trial as clinically indicated. Patients may also undergo bone scans on study and may undergo biopsies throughout the study as clinically indicated.
  Interventions: Drug: Binimetinib; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Echocardiography Test; Drug: Fluorouracil; Drug: Leucovorin Calcium; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Binimetinib — Given PO
  Other Names: ARRY 162; ARRY 438162; ARRY-162; ARRY-438162; ARRY162; ARRY438162; MEK 162; MEK-162; MEK162; Mektovi
  Arms: Arm 2 (binimetinib, mFOLFOX6)
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
  Arms: Arm 2 (binimetinib, mFOLFOX6)
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Drug: Leucovorin Calcium — Given IV
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
  Arms: Arm 2 (binimetinib, mFOLFOX6)
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; Elplat; JM 83; JM-83; JM83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; RP54780; SR 96669; SR-96669; SR96669

SUMMARY:
This phase II ComboMATCH treatment trial compares the usual treatment of modified leucovorin, fluorouracil and oxaliplatin (mFOLFOX6) chemotherapy to using binimetinib plus mFOLFOX6 chemotherapy to shrink tumors in patients with biliary tract cancers that have spread to other places in the body (advanced) and had progression of cancer after previous treatments (2nd line setting). Fluorouracil is in a class of medications called antimetabolites. It works by slowing or stopping the growth of cancer cells in the body. Oxaliplatin is in a class of medications called platinum-containing antineoplastic agents. It works by killing tumor cells. Leucovorin may help the other drugs in the mFOLFOX6 chemotherapy regimen work better by making tumor cells more sensitive to the drugs. Binimetinib is in a class of medications called kinase inhibitors. It works by blocking the action of the abnormal protein that signals tumor cells to multiply. This helps to stop or slow the spread of tumor cells. Giving binimetinib in combination with mFOLFOX6 chemotherapy may be effective in shrinking or stabilizing advanced biliary tract cancers in the 2nd line setting.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether binimetinib and mFOLFOX6 combination therapy improves overall survival (OS) compared to mFOLFOX6 alone in patients with advanced/recurrent biliary tract cancer (BTC) and with alterations in RAS/RAF/MEK/ERK pathway, who have progressed on one prior line of therapy.

SECONDARY OBJECTIVES:

I. To determine whether binimetinib and mFOLFOX6 combination therapy improves objective response rate (ORR) compared to FOLFOX alone.

II. To determine if clinical outcomes including progression free survival (PFS), duration of response (DOR), and disease control rate (DCR) are improved with combination treatment of binimetinib and mFOLFOX6 compared to FOLFOX alone in patients with advanced/recurrent BTC and with alterations in RAS/RAF/MEK/ERK pathway who have progression on one prior line of therapy.

III. Toxicity and tolerability will be evaluated within and between the two treatment arms, where frequency, type, and severity of adverse events will be assessed per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version (v)5.0.

IV. Collect tissue and provide it to the ComboMATCH Registration Protocol to assess concordance between the diagnostic tumor mutation profile generated by the Designated Laboratories, the pre-treatment biopsy mutation profile, and the pre-treatment circulating tumor deoxyribonucleic acid (ctDNA) mutation profile from plasma, as described in ComboMATCH Registration Protocol.

EXPLORATORY OBJECTIVES:

I. Generate a prognostic model of MAPK mutations for this patient population using clinical, laboratory and molecular features of their disease and clinical outcome to validate on future samples.

II. Correlation of outcome with albumin. III. Assess the correlation between the presence of MAPK pathway mutations and activity of addition of binimetinib therapy to standard 2nd line chemotherapy.

IV. Conduct whole-exome sequencing and ribonucleic acid (RNA)-sequencing at baseline, and on optional biopsy upon progression to assess determinants of response and resistance.

V. Explore changes in plasma MAPK mutations allelic burden and other molecular findings at baseline and upon progression using ctDNA and correlate changes with clinical activity, disease course as well as response/resistance to therapy.

VI. Evaluate if our machine learning algorithm for RAS/RAF/MEK/ERK pathway mutations correlates with detection of mutations as well as prediction of outcomes from samples obtained in this study.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM 1: Patients receive leucovorin intravenously (IV) over 2 hours and oxaliplatin IV over 2 hours on day 1, and fluorouracil IV over 46-48 hours on days 1-2. Cycles repeat every 14 days in the absence of disease progression or unacceptable toxicity. Patients undergo collection of blood during screening and on study, and undergo computed tomography (CT) with contrast, magnetic resonance imaging (MRI), or fludeoxyglucose F-18 positron emission tomography (FDG-PET) throughout the trial as clinically indicated. Patients may also undergo bone scans on study and may undergo biopsies throughout the study as clinically indicated.

ARM 2: Patients receive binimetinib orally (PO) on days 1-14, and leucovorin IV, oxaliplatin IV, and fluorouracil IV as in Arm 1. Cycles repeat every 14 days in the absence of disease progression or unacceptable toxicity. Patients undergo echocardiogram (ECHO) or multigated acquisition scan (MUGA) and collection of blood during screening and on study, and undergo CT with contrast, MRI, or FDG-PET throughout the trial as clinically indicated. Patients may also undergo bone scans on study and may undergo biopsies throughout the study as clinically indicated.

After completion of study treatment, patients are followed up every 8 weeks until disease progression, thereafter patients are followed for survival every 4 months for up to 5 years following registration.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have enrolled onto EAY191 and must have been given a treatment assignment to ComboMATCH to EAY191-A6 based on the presence of an actionable mutation as defined in EAY191
* GENERAL COMBOMATCH EAY191:
* Patients must be registered to the ComboMATCH Registration Protocol (EAY191)
* Patients must have RAS/RAF/MEK/ERK mutations as determined by the ComboMATCH screening assessment
* Patients must not have BRAF V600E as determined by the ComboMATCH screening assessment
* Patients must have disease that can be safely biopsied and agree to a pre-treatment biopsy or have archival tissue available from within 12 months prior to registration on the ComboMATCH Registration Trial (EAY191).
* Please note the current actionable marker of interest (aMOI)/actionable alteration list for this treatment trial can be found on the Cancer Trials Support Unit (CTSU) website
* Please note novel/Dynamic aMOI can be submitted for review per the process described in the ComboMATCH Registration Protocol
* EAY191-A6 REGISTRATION:
* Participants must have histologically confirmed BTC (intrahepatic cholangiocarcinoma [IHC], extrahepatic cholangiocarcinoma [EHC] or gallbladder cancer [GBC]) that is unresectable or recurrent with a confirmed RAS/RAF/MEK/ERK pathway mutation via any Clinical Laboratory Improvement Act (CLIA)-certified method. BRAFV600E mutations are not eligible due to other ongoing/upcoming studies in this disease cohort
* Tumor tissue must be available:

  * Adequate archival tumor specimen (obtained within 12 months of EAY191 registration which has not had a Response Evaluation Criteria in Solid Tumors (RECIST) response, complete response (CR) or partial response (PR), to any intervening therapy after collection of the tissue) must be available with formalin-fixed paraffin-embedded tumor tissue (blocks or slides) OR
  * Consent to a new tumor tissue biopsy which is not a representative target lesion. This lesion must be amenable to a minimal risk image-guided or direct vision biopsy

    * A new biopsy is preferred but is not required for enrollment in EAY191-A6 if sufficient archival tissue is available as described above.
* Measurable disease per RECIST 1.1 Of note, in the case when a baseline biopsy is done after scans are obtained, a lesion separate from one that is biopsied needs to be measurable per RECIST 1.1. All radiologic studies must be performed within 28 days prior to registration
* Progression of disease on gemcitabine based first-line regimen (i.e. only one prior line of therapy is permitted)
* No systemic anti-cancer therapy within 4 weeks of registration to EAY191-A6
* No prior MEK inhibitor therapy
* No prior history of treatment with a direct and specific inhibitor of KRAS
* Patients who only received radio-sensitizing chemotherapy with fluorouracil (5-FU) or capecitabine are eligible, but need to have received and failed first-line systemic chemotherapy upon recurrence. Peri-operative systemic 5-FU/capecitabine and/or oxaliplatin, is allowed if it's been more than 12 months of registration to EAY191-A6
* No major surgery within 4 weeks (excluding placement of vascular access) of registration to EAY191-A6
* No minor surgery within 2 weeks of registration to EAY191-A6
* No palliative radiotherapy within 1 week of registration to EAY191-A6
* Not pregnant and not nursing, because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown

  * Therefore, for women of childbearing potential only, a negative pregnancy test done =< 14 days prior to registration is required
  * Adequate contraception is needed for at least 30 days after the last dose of binimetinib and breastfeeding should be discontinued for at least 3 days after the last dose of binimetinib. For FOLFOX regimen, 9 months is recommended for contraception after last dose of oxaliplatin for females of childbearing potential and 6 months for males
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Absolute neutrophil count (ANC) >= 1,000/mm^3, no growth factor within 14 days of 1st dose
* Platelet count >= 75,000/mm^3
* Creatinine < 1.6 x upper limit of normal (ULN) OR
* Calculated (Calc.) creatinine clearance >= 50 mL/min, as calculated by the Cockcroft-Gault formula
* Total bilirubin =< 2.0 x upper limit of normal (ULN); Patients with Gilbert syndrome may enroll if < 3.0 x ULN
* Aspartate aminotransferase (AST) /alanine aminotransferase (ALT) =< 5.0 x upper limit of normal (ULN)
* Hemoglobin >= 8 g/dL, no transfusion within 7 days of 1st dose
* Creatine phosphokinase =< 2.5 x ULN
* High blood pressure more than 160/90 despite treatment are ineligible
* No history of interstitial lung disease. No history of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* Patients should not have history of bowel perforation or intestinal fistulas in the last 6 months
* Patients with the inability to swallow oral medications or impaired gastrointestinal absorption due to gastrectomy or active inflammatory bowel disease are ineligible
* Must have adequate cardiac function with left ventricular ejection fraction >= 50% by echocardiography (ECHO) or multiple-gated acquisition (MUGA) scan. Patients with congenital long QT syndrome are not permitted
* No history of prolonged QTc or at risk for prolonged QTc due to any reason (for example, concomitant medications during or before chemotherapy that may increase the risk of prolonged QTc), uncontrolled congestive heart failure, prior history of class III/ IV cardiac disease (New York Heart Association [NYHA]), myocardial infarction within the last 6 months, unstable arrhythmias, unstable angina or severe obstructive pulmonary disease
* No active skin disorder that has required systemic therapy within the past 1 year
* No history of rhabdomyolysis
* No concurrent ocular disorders, including:

  * Patients with history of glaucoma, history of retinal vein occlusion (RVO), predisposing factors for RVO, including but not limited to uncontrolled hypertension, uncontrolled diabetes
  * Patients with history of retinal pathology or evidence of visible retinal pathology that is considered a risk factor for RVO, intraocular pressure > 21 mm Hg as measured by tonometry, or other significant ocular pathology, such as anatomical abnormalities that increase the risk for RVO
  * Patients with a history of corneal erosion (instability of corneal epithelium), corneal degeneration, active or recurrent keratitis, and other forms of serious ocular surface inflammatory conditions
  * Patients with known or at risk for retinopathies, uveitis or retinal vein occlusion
* No patients with a history of hypersensitivity to any of the inactive ingredients in binimetinib, nor known severe allergic reactions or hypersensitivity of 5-FU, leucovorin (LV) or oxaliplatin will be allowed to participate in this study for safety concerns
* No other medical condition (e.g. cardiac, gastrointestinal, pulmonary, psychiatric, neurological, genetic, etc.) that in the opinion of the investigator would places the subject at unacceptably high risk for toxicity
* No prior allogeneic stem cell or solid organ transplantation
* Central nervous system (CNS) metastases must have been treated with local therapy (surgery, radiation, ablation) with systemic steroids tapered to a physiologic dose (10 mg or prednisone equivalent or less)
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients must not have grade 2 neuropathy or greater, within 14 days prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-02-09 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From randomization to the time of death due to any cause, assessed up to 30 months
  The primary efficacy analysis will be to compare the OS distributions between those treated with modified leucovorin, fluorouracil and oxaliplatin (mFOLFOX6) and binimetinib versus (vs.) mFOLFOX6. Despite being a randomized phase II trial, we will utilize an intent to treat approach such that patients will be analyzed based on the treatment arm to which they were randomized. As defined above, OS will be compared between the two treatment arms using Kaplan-Meier methods. The hazard ratio, median OS, and estimated OS rates at 6, 12, 18, 24, and 30 months will be estimated along with corresponding 95% confidence intervals. Anticipating that the treatment arms will be balanced in terms of the potential confounders reflect in the stratification factors, a log-rank test will be used to compare the OS distributions between the two treatment arms in this cohort.

SECONDARY OUTCOMES:
Objective response | Up to 5 years
  Objective response by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 criteria will be estimated using objective response rate (ORR) where ORR is defined as the number of evaluable patients achieving a response (partial response [PR] or complete response [CR] per RECIST v1.1) during treatment with study therapy divided by the total number of evaluable patients. Rates of response will be compared across arms using a Chi-Square Test for Proportion. Point estimates will be generated for objective response rates within each arm along with 95% confidence intervals using the Clopper-Pearson method.
Progression free survival (PFS) | From study entry to the first of either disease progression or death from any cause, assessed up to 5 years
  Disease progression will be determined based on RECIST 1.1 criteria. PFS will be estimated using the Kaplan-Meier method. The median PFS and 95% confidence interval will be reported. Patients will be censored at the last disease assessment date.
Duration of response (DoR) | Up to 5 years
  Defined for all evaluable patients who have achieved an objective response as the date at which the patient's earliest best objective status is first noted to be either a CR or PR to the earliest date progression is documented, or death if no prior evidence of disease progression. The distribution of DoR will be estimated using the method of Kaplan-Meier.
Clinical benefit | Up to 5 years
  Defined as achieving CR, PR, or stable disease (SD) for at least 4 months while on treatment. Disease status will be assessed using RECIST v. 1.1 criteria. Clinical benefit rate (CBR) will be calculated as the proportion of evaluable patients who achieve clinical benefit. The final CBR point estimate and corresponding 95% confidence interval calculated using Clopper-Pearson method.
Incidence of adverse events | Up to 5 years
  Patients will be evaluated for adverse events using the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events version 5.0. Summary statistics (e.g., mean, median, standard deviation) and frequency tables will be used to describe the distributions of adverse events. Rates of adverse events occurring in the treatment arm will be compared to the control arm with chi-squared tests (or suitable alternative) used for comparisons where applicable. Tolerability will also be evaluated, summarizing rates of dose delays or modifications, reasons patients end treatment, and time to end of active treatment.

OTHER OUTCOMES:
Prognostic model/scoring system | Up to 5 years
  Defined as presence of peritoneal disease/locally advanced disease/metastatic disease, Eastern Cooperative Oncology Group (ECOG) performance status, CA19.9 level. Will fit multivariate Cox regression models including MAPK mutation status, presence of peritoneal disease/locally advance disease/metastatic disease, ECOG performance status, and CA19-9 level, stratified by treatment arm. We will calculate C-statistics with 5-fold cross-validation
Albumin | Up to 5 years
  Will correlate outcome with albumin.
Presence of MAPK pathway mutations | Up to 5 years
  Will correlate with activity of addition of binimetinib therapy to standard 2nd line chemotherapy.
Activity of addition of binimetinib therapy to standard 2nd line chemotherapy | Up to 5 years
  Will correlate with presence of MAPK pathway mutations.
Whole-exome sequencing and ribonucleic acid (RNA)-sequencing | Up to 5 years
  Will be used to assess determinants of response and resistance. Concordance of diagnostic tumor mutation profile generated by the Designated Laboratory, the pre-treatment biopsy mutation profile, and the pre-treatment circulating tumor deoxyribonucleic acid (ctDNA) mutation profile will be assessed. Details are provided in the statistical plan of the ComboMATCH Registration Protocol.
Changes in plasma MAPK mutations allelic burden and other molecular findings | Up to 5 years
  Will correlate changes with clinical activity, disease course as well as response/resistance to therapy.
Detection of mutations as well as prediction of outcomes | Up to 5 years
  Will evaluate if our machine learning algorithm for RAS/RAF/MEK/ERK pathway mutations correlates with detection of mutations as well as prediction of outcomes from samples obtained in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Ardaman Shergill, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (209):
- United States (209):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Presbyterian Intercommunity Hospital, Whittier, California
  - UM Sylvester Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - The Queen's Medical Center - West Oahu, ‘Ewa Beach, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - UPMC Western Maryland, Cumberland, Maryland
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - University of Michigan - Brighton Center for Specialty Care, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Miami Valley Hospital South, Centerville, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - UPMC Altoona, Altoona, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - UPMC Hillman Cancer Center - Monroeville, Monroeville, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - MD Anderson in The Woodlands, Conroe, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Valley Medical Center, Renton, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - ThedaCare Cancer Care - Berlin, Berlin, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Saint Luke's South Shore, Cudahy, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - ThedaCare Regional Medical Center - Neenah, Neenah, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm